CLINICAL TRIAL: NCT03901508
Title: A Single Session of a-tDCS Improves Lower Limb Endurance for 30 Minutes in Healthy Subjects
Brief Title: A Single Session of tDCS (Transcranial Direct Current Stimulation) Improves Endurance for 30 Minutes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2017/29
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Athlete; Healthy
Keywords: tDCS; Athlete; Isokinetic; Strength; Endurance
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, sham-controlled, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The device is preprogrammed by a third party non participating in any element in the study. They then chose (using opaque envelopes) the treatment code for each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): Subjects will receive 20min anodal tDCS
  Interventions: Device: TDCS
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of Sham anodal tDCS
  Interventions: Device: TDCS

INTERVENTIONS:
Device: TDCS — 20 minutes, 2 electrodes (C3/FP2)
  Other Names: Non invasive brain stimulation

SUMMARY:
Healthy recreational athletes will undergo a session of anodal tDCS (transcranial direct current stimulation) or sham tDCS.

The primary outcome is an isokinetic evaluation of their hamstrings' and quadriceps' strength before and after each session

DETAILED DESCRIPTION:
Healthy recreational athletes will be recruited through social media and advertisements.

Each subject came to the Liege University Hospitals' isokinetic lab. Each session began with strapping the subjet into the isokinetic machine, making sure that all the settings were adapted to the subject. Then, each subject underwent a concentric and eccentric isokinetic test of their lower limbs (dominant or non-dominant side depending on their group). Subjects then received either anodal tDCS, of sham tDCS. Neither the evaluator or the subject knew which they were receiving. Immediately following tDCS, there was a another isokinetic test, and 30 minutes after the second test, a subjects underwent a third test.

ELIGIBILITY:
Inclusion Criteria:

* Between 3 and 5 hours of sport a week
* Right handed and footed

Exclusion Criteria:

* One on the TSST (in high and relatively high risk sections)
* Previous neurological or orthopedic pathologies affecting limbs

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Isokinetic Peak Strength | Changes between prior to tDCS, immediately following tDCS and 30 minutes after tDCS
  Concentric and Eccentric Peak Strength is measured in hamstrings and quadriceps at 60°/s using an isokinetic dynamometer
Isokinetic Work | Changes between prior to tDCS, immediately following tDCS and 30 minutes after tDCS
  Concentric and Eccentric Work is measured in hamstrings and quadriceps at 60°/s using an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bornheim, Msc, Principal Investigator — Liege University Hospital
Locations (1):
- Liege Univeristy Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No